CLINICAL TRIAL: NCT01950052
Title: Randomised Controlled Trial to Study the Effects of Preoperative Very Low Calorie Diet on Wound Healing in Morbidly Obese Patients Undergoing Bariatric Surgery
Brief Title: Pre-operative Diet: Effect of Wound Healing After Bariatric Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KCH12-109
Record Dates: First submitted 2013-09-18; First posted 2013-09-25 (Estimated); Last update posted 2016-06-09 (Estimated); Status verified 2016-02

CONDITIONS: Obese
Keywords: VLCD; Low calorie diet; very low calorie diet; pre-operative diet; liver shrinking diet; bariatric surgery; gastric bypass
MeSH Terms: conditions — Obesity | interventions — Diet

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): No special diet, patients will continue with a normal diet
- Diet group (Experimental): Pre-operative liver shrinking diet of 800 Kcal diet is administered for 4 weeks
  Interventions: Dietary Supplement: Diet group 800 Kcal diet

INTERVENTIONS:
Dietary Supplement: Diet group 800 Kcal diet — Pre-operative liver shrinking diet of 800 kcal is administered for 4 weeks
  Other Names: VLCD
  Arms: Diet group

SUMMARY:
This study is a randomised control trial comparing the effects of a pre-operative very low calorie diet (VLCD) on wound healing in the morbidly obese patients undergoing bariatric surgery.

The benefits and disadvantages of a very low calorie pre-operative diet are not clear. Some centres ask their patients to take a VLCD 2-6 weeks before bariatric surgery with the aim of shrinking the liver to make surgery easier. Studies have shown that after this diet the liver does shrink and therefore operating may be easier but this did not necessary translate into significant lesser operative times. The effects of operating during a catabolic phase have not been evaluated. Theoretically a low calorie diet before surgery is similar to starving a patient and can potentially create a state of malnutrition. This is rarely advisable before surgery and can lead to poor wound healing and poor healing of bowel anastomosis.

This study will ascertain if there is any difference in wound healing rates in these morbidly obese patients (BMI>40kg/m2)undergoing a Laparoscopic Roux en Y gastric by pass in groups who have taken the preoperative diet compared to those who were not on a special diet. Skin wounds will be evaluated. This will potentially reflect the general state of healing of the patient which includes the healing of bowel anastomosis. Surrogate markers will be employed to evaluate the pre-morbid nutritional state, effectiveness of dieting, subsequent wound healing (collagen production, markers for the different aspects of wound healing) and impact on liver cell death .This study will be able to tell us how safe this calorie deficient diet is in these morbidly obese patients before surgery.

DETAILED DESCRIPTION:
Study Design:

Prospective single blinded randomised controlled study

Null hypothesis: There is no difference in wound healing between patients on a very low calorie diet and those not on a diet prior to a Laparoscopic Roux en Y gastric bypass (LRYGB)

Participants:

All patients referred to King's College Hospital for weight loss surgery who are morbidly obese (BMI>40) who undergo LRYGB will be eligible. All patients undergo an introductory group education session after which they are counselled one to one where the patient and the clinician decide on the most appropriate bariatric procedure. Only those who will undergo a laparoscopic roux en y gastric bypass will be offered the opportunity to participate in the study by a member of the research team. The study is open to all irrespective of age, sex, ethnicity and religion.

Written information will be given in the appropriate language.

Interventions:

Diet:

Patients who meet the eligibility criteria will be placed in 2 broad groups based on whether they smoke or not. In each group, patients will be randomly chosen in two subgroups:

Group I:taking the pre operative diet Group II:no special diet. A preoperative, low energy diet will be used for 4 weeks. The diet contains 3 pints of semiskimmed milk. This is equivalent to 1704 ml and provides a total intake of 800kcal, 82 g carbohydrate, 61 g protein and 30g fat in a day. Each patient will also take multivitamin and mineral supplementation. This will further be supplemented with a minimum of 2 litres of energy free liquids (water, diet fizzy drinks, mineral water, black tea / coffee or squash (no added sugar)) per day. The longterm safety and success of VLCD has been demonstrated.It does cause shrinkage of the liver and can decrease the patients weight prior to surgery.

Data collection:

Patient characteristics and medical history will be taken

Pre diet, post diet and prior to surgery:

1. Anthropometric measurements:

   Height, Weight, BMI, Hip:Waist ratio
2. Routine prediet blood tests and for routine preoperative evaluation:

   This includes full blood count,Lipid profile,Renal profile,Bone profile,Liver Function Tests
3. Serum CK 18 (M30 and M65) levels before and after the diet, which is a marker of liver apoptosis.
4. Imaging:

   1. Dual-energy X-ray absorptiometry (DEXA) scan - body composition (prediet,post diet and at 3 months)
   2. Ultrasound before and after the diet:

   The length and breadth of the liver will be measured, which will allow an estimate of the cross-section of the liver at a well defined constant point on each patient
5. Two punch biopsies (4mm) from the abdominal wall where the patient is likely to have a laparoscopic port, before start of the diet

Per operatively:

* Elliptical excision of skin of the operating ports during the operation
* Operative difficulty score assessed by blinded surgeon and independent observer

Post operatively:

Follow up:

Patient will be followed at 1 week, 8 weeks, 3 months and then will continue to be followed according to our usual bariatric protocol.

Wound Healing Assessment:

1. Examine all wounds and define presence of wound infection
2. Two 4 mm punch biopsies of one of the healing wounds will be taken under local anaesthesia, at 7 days and 90 days postoperatively

ELIGIBILITY:
Inclusion Criteria:

* Patients who have given written informed consent
* Patients who are able to understand and comply with protocol requirements
* Patients 18-70 years old
* Patients scheduled for Laparoscopic Roux En Y Gastric Bypass
* Patients with BMI > 40 and < 60

Exclusion Criteria:

* Unable or unwilling to give an informed written consent
* Cognitive impairment or mental retardation
* Patient who do not understand or follow protocol requirements
* Severe hepatic impairment or portal hypertension
* Pregnancy and lactation
* Diabetes
* Pre-existing chronic inflammatory disease
* Overt psychosis
* Porphyria
* Advanced renal disease
* Acute cerebrovascular or cardiovascular disease
* Patients with alcohol or drug addiction
* Patients taking medication known to impact wound healing (eg glucocorticosteroids, chemotherapy, immunosuppressant)
* Patients who lose less than 5% of body weight after 4 weeks of the diet

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-11; Primary Completion 2016-11 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Collagen 1/3 ratio after diet and surgery | 7 days following surgery
  Special immunostains for collagen 1 and 3 will be utilised and their ratio will be calculated by an independent blinded operator

SECONDARY OUTCOMES:
Is there any difference in wound healing between patients undergoing aggressive calorie restriction and those without a dietary intervention prior to bariatric surgery? | 7 days following surgery
  Changes in elastin,fibrinogen,myofibroblasts and angiogenesis (formation of new blood vessels) will be evaluated using special immunostains
Change in body composition between control group and patients with diet | At one moth after the diet and 3 months following surgery
  DEXA scans will be performed for body composition analysis

OTHER OUTCOMES:
Is there any difference in liver volume and fibrosis between control group and patients with diet? | Outcomes will measured at 1 month compared to baseline values

CONTACTS AND LOCATIONS:
Overall Officials: Ameet G Patel, MS FRCS, Principal Investigator — King's College Hospital NHS Trust
Locations (1):
- King's College Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided